CLINICAL TRIAL: NCT05518058
Title: Effect of Electromyography Triggered Functional Electrical Stimulation on Stroke Patients
Brief Title: Electromyography Triggered Functional Electrical Stimulation on Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, Hend Elsharkawy, Assistant lecturer, Delta University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Delta 2022
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2022-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Experimental): strengthening exercises program plus balance exercises program
  Interventions: Other: device and exercises
- Study group (Experimental): strengthening exercises program plus balance exercises program conducted with EMG triggered FES
  Interventions: Other: device and exercises

INTERVENTIONS:
Other: device and exercises — strengthening exercises plus balance training program conducted with type of functional electrical stimulation for muscles
  Other Names: therapeutic exercises program / EMG triggered FES device

SUMMARY:
my study aims to apply treatment program for postural instability in stroke patients.

DETAILED DESCRIPTION:
my study include two groups: first group receive physical therapy exercise program followed by balance exercise program.

the second group receive the same physical therapy exercise program followed by balance exercise program conducted with electromyography triggered functional electrical stimulation

ELIGIBILITY:
Inclusion Criteria:

* stroke patients
* normal body mass index
* mild spasticity

Exclusion Criteria:

* musculoskeletal deformities
* cognitive abnormalities
* cardiovascular diseases

Ages: 45 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Postural stability | 2 months
  biodex balance system

SECONDARY OUTCOMES:
dynamic balance | 2 months
  timed up and go test

CONTACTS AND LOCATIONS:
Locations (1):
- Hend Elsharkawy, Damietta, Texas, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: after 12 months from publication